CLINICAL TRIAL: NCT00187395
Title: Control of Hypertension in Pregnancy Study: A Pilot Trial
Brief Title: CHIPS (Control of Hypertension in Pregnancy Study): A Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCT- 59755; ISRCTN57277508
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2005-09

CONDITIONS: Transient Hypertension, Pregnancy
Keywords: hypertension; blood pressure; pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension

INTERVENTIONS:
Procedure: Randomized to either a 'less tight' group or a 'tight' group

SUMMARY:
Prior to undertaking CHIPS which will be a large and difficult trial, we believe we need to first determine whether clinicians will comply with the interventions of 'less tight' and 'tight' control of dBP, and whether the interventions will result in differences in mean dBP between groups. A pilot will also allow us to confirm the ability of centres to identify eligible women and the willingness of women to join CHIPS.

DETAILED DESCRIPTION:
To determine whether 'less tight' control of mild-moderate non-proteinuric maternal hypertension, aiming for a diastolic blood pressure (dBP) of 100mmHg, can decrease the risks of adverse perinatal outcome without increasing maternal risk compared with 'tight' control, aiming for a dBP of 85mmHg.

ELIGIBILITY:
Inclusion Criteria:

* dBP 90-109mmHg due to pre-existing or gestational hypertension; live fetus(es); and 20-33+6 weeks.

Exclusion Criteria:

* dBP consistently < 85mmHg by home BP monitoring; severe systolic hypertension; proteinuria; contraindication to either arm of the trial or to prolongation of pregnancy; or known lethal/major fetal anomaly.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132
Dates: Start 2003-04; Study Completion 2005-12

PRIMARY OUTCOMES:
Mean dBP at 28, 32 and 36 weeks gestation

SECONDARY OUTCOMES:
Clinician compliance with treatment protocols; women's satisfaction with care.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Magee, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Maternal Infant and Reproducting Health Research Unit - CHIPS Data Coordinating Centre, Toronto, Ontario, Canada